CLINICAL TRIAL: NCT04869085
Title: The Use of a Digital Application for Reporting Pain and Pain Management in Home Hospice
Acronym: ePainSupport
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Masako Mayahara, Associate Professor and Associate Chairperson, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19111205-IRB01; 5R21NR018952 (NIH); 310245 (Other: Rush University); 310244 (Other: Rush University); 310243 (Other: Rush Univesrity)
Record Dates: First submitted 2021-03-19; First posted 2021-05-03 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Pain
Keywords: Pain, Pain management, Analgesics, Adherence; Hospice, End-of-Life Care; Caregiver; m-Health, digital interventions
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Data Collectors will be blinded to the intervention. Study participants will be asked to not disclose their treatment condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- e-PainSupport Condition (Experimental): e-PainSupport is a self-administered, digital pain application. Over the course of the two weeks, caregivers and patients will record the severity of patient's pain and how much pain medicine they use to control patient's pain in the e-PainSupport application.
  Interventions: Behavioral: e-PainSupport
- Standard Care Condition (No Intervention): Patients and caregivers will be given a paper copy of the same list of resources for pain management included in the Education Module of the e-PainSupport condition at baseline.

INTERVENTIONS:
Behavioral: e-PainSupport — Patients and caregivers assigned to the e-PainSupport condition will download the app on their own device, or they will be given a project tablet with wireless capability if they do not have their own device. All receive specific training for the intervention. They will also receive a hardcopy of the e-PainSupport manual and a trouble-shooting guide. Contact information will be provided in the app and on paper for technical problems. Caregivers complete Education Module, and patients may complete it. Caregiver or patient will fill out Pain Report daily. Pain Summary for Nurses is an automatically generated graphic summary of patients' Pain Reports over time. Nurses have access to this information during the time the patients and caregivers use e-PainSupport.
  Arms: e-PainSupport Condition

SUMMARY:
Poor adherence to pain management and high pain intensity associated with serious, advanced illness is a major public health concern. This randomized clinical trial will test the efficacy of a newly enhanced digital pain and pain management application (e-PainSupport) for use in a home hospice setting. The e-PainSupport application delivers an education module about pain management to patients and caregivers, expedites pain reporting to nurses, and facilitates adherence to pain management. The overall goal of the e-PainSupport application is to improve pain management and reduce patient pain intensity in the home hospice setting.

DETAILED DESCRIPTION:
High pain intensity is a common symptom experienced by patients with serious advanced illness. However, pain management for patients in home hospice is less than optimal. Impediments to improving pain intensity are poor adherence to pain management regimen due in part to caregiver lack of knowledge (a barrier to reporting pain and using analgesics) and lack of self-efficacy (confidence) in administering analgesics. Digital applications may facilitate pain management by: (1) delivering education to increase knowledge and self-efficacy, (2) expediting pain reporting to nurses, and (3) improving adherence to pain management. e-PainSupport is a self-administered, digital pain management application developed in collaboration with hospice nurses and caregivers. It is directly linked to a patient's medical record and enhanced by an evidence-based educational module. It has three elements: (a) Educational Module, (b) Patient Pain Record, and (c) Pain Summary for Nurses. The purpose of this study is to test the effects of e-PainSupport on home hospice patient pain intensity when used by patients, caregivers and nurses. Participants (132 triads of patient, caregiver, and the hospice nurse assigned to the patient will be recruited from one large Midwest hospice agency. Patient and caregiver outcomes will be assessed at baseline and 2 weeks post baseline. Data will be analyzed with multi-level modeling. Post-intervention semi-structured interviews will be conducted with nurses who provided care to patients in the e-PainSupport condition. Qualitative content analysis will be used to identify themes related to perceived practice changes after using e-PainSupport. e-PainSupport has potential as a useful tool to advance home hospice care by enhancing the quality of caregiver pain management, facilitating nurse-patient communication, and improving management of patient pain intensity.

ELIGIBILITY:
Inclusion criteria (patient)

* prior enrollment of their hospice nurse
* receives analgesics for pain
* speaks and reads English
* age 18 or older
* has a primary informal caregiver who is available for the 2 weeks of the study
* expected survival of at least 2 weeks
* can verbalize pain.

Inclusion criteria (caregiver)

* speaks and reads English
* age 18 or older
* cares for an enrolled patient
* available for the 2 weeks of the study.

Inclusion criteria (nurses participating in the RTC)

* registered nurse (RN)
* provides direct care to patients
* has not had a prior patient enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Minimally important clinical change in pain intensity (at least 10 percent change on the pain intensity scale) | Baseline
  Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity-Short Form 3a v1.0 v3 items: worst pain and average pain in past 7 days, and current pain, scored from 1 = no pain, 2= mild, 3 = moderate, 4= severe, 5 = very severe pain, summed for a range of 3 to 15. Higher scores indicates higher pain intensity.
Minimally important clinical change in pain intensity (at least 10 percent change on the pain intensity scale) | 2-weeks post baseline
  Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity-Short Form 3a v1.0: 3 items: worst pain and average pain in past 7 days, and current pain, scored from 1 = no pain, 2= mild, 3 = moderate, 4= severe, 5 = very severe pain, summed for a range of 3 to 15. Higher scores indicates higher pain intensity.

SECONDARY OUTCOMES:
Change in the continuous score of the pain intensity scale | Baseline
  Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity-Short Form 3a v1.0: 3 items: worst pain and average pain in past 7 days, and current pain, scored from 1 = no pain, 2= mild, 3 = moderate, 4= severe, 5 = very severe pain, summed for a range of 3 to 15. Higher scores indicates higher pain intensity.
Change in the continuous score of the pain intensity scale | 2-weeks post baseline
  Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity-Short Form 3a v1.0. 3items: worst pain and average pain in past 7 days, and current pain, scored from 1 = no pain, 2= mild, 3 = moderate, 4= severe, 5 = very severe pain, summed for a range of 3 to 15. Higher scores indicates higher pain intensity.

OTHER OUTCOMES:
Self-Efficacy | Baseline
  Chronic Pain Self-Efficacy Scale: Self-efficacy for pain management subscale measures confidence in managing pain, 5 items on 10-point Likert scale anchored on the ends by 10=very uncertain and 100=very certain. The score ranges from 50 to 500. Higher scores indicate higher perceived self efficacy.
Self-Efficacy | 2-weeks post baseline
  Chronic Pain Self-Efficacy Scale: Self-efficacy for pain management subscale measures confidence in managing pain, 5 items on a 10-point Likert scale anchored on the ends by 10=very uncertain and 100=very certain. The score ranges from 50 to 500. Higher scores indicate higher perceived self efficacy.
Adherence to pain management | Baseline
  Morisky Medication Adherence Scale-4 item version: Measures medication adherence, 4 items on a five-point Likert scale. Patients answer yes or no to questions (e.g., Do you sometimes forget to take your pain medication?).Each "yes" answer is scored as 1.The score ranges from 0 to 4. Lower score indicates better adherence.
Adherence to pain management | 2-weeks post baseline
  Morisky Medication Adherence Scale-4 item version : Measures medication adherence, 4 items on a five-point Likert scale. Patients answer yes or no to questions (e.g., Do you sometimes forget to take your pain medication?). Each "yes" answer is scored as 1. The score ranges from 0 to 4. Lower score indicates better adherence.
Knowledge | Baseline
  Barriers Questionnaire II measures 8 knowledge barriers about reporting pain and using analgesics, with four subscales (physiological effects, 12 items; fatalism, 3 items; communication, 6 items; and harmful effects, 6 items (total 27 items) on a 6-point scale (0 = don't agree, 5 = agree very much), items averaged (range 0 to 5). The score ranges from 0-135. Higher scores indicate stronger barriers.
Knowledge | 2-weeks post baseline
  Barriers Questionnaire II (BQ-II) measures 8 knowledge barriers about reporting pain and using analgesics, with four subscales (physiological effects, 12 items; fatalism, 3 items; communication, 6 items; and harmful effects, 6 items (total 27 items), 6-point scale (0 = don't agree, 5 = agree very much), items averaged (range 0 to 5).The score ranges from 0-135. Higher scores indicate stronger barriers.

CONTACTS AND LOCATIONS:
Overall Officials: Masako Mayahara, PhD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keefe FJ, Ahles TA, Porter LS, Sutton LM, McBride CM, Pope MS, McKinstry ET, Furstenberg CP, Dalton J, Baucom DH. The self-efficacy of family caregivers for helping cancer patients manage pain at end-of-life. Pain. 2003 May;103(1-2):157-62. doi: 10.1016/s0304-3959(02)00448-7. PMID 12749970
- [Background] Dworkin RH, Turk DC, McDermott MP, Peirce-Sandner S, Burke LB, Cowan P, Farrar JT, Hertz S, Raja SN, Rappaport BA, Rauschkolb C, Sampaio C. Interpreting the clinical importance of group differences in chronic pain clinical trials: IMMPACT recommendations. Pain. 2009 Dec;146(3):238-244. doi: 10.1016/j.pain.2009.08.019. PMID 19836888
- [Background] Borneman T, Koczywas M, Sun V, Piper BF, Smith-Idell C, Laroya B, Uman G, Ferrell B. Effectiveness of a clinical intervention to eliminate barriers to pain and fatigue management in oncology. J Palliat Med. 2011 Feb;14(2):197-205. doi: 10.1089/jpm.2010.0268. Epub 2011 Jan 27. PMID 21271872
- [Background] Irani E, Hirschman KB, Cacchione PZ, Bowles KH. How home health nurses plan their work schedules: A qualitative descriptive study. J Clin Nurs. 2018 Nov;27(21-22):4066-4076. doi: 10.1111/jocn.14548. Epub 2018 Jul 23. PMID 29893442
- [Result] Kehl KA, Kowalkowski JA. A systematic review of the prevalence of signs of impending death and symptoms in the last 2 weeks of life. Am J Hosp Palliat Care. 2013 Sep;30(6):601-16. doi: 10.1177/1049909112468222. Epub 2012 Dec 12. PMID 23236090
- [Result] Singer AE, Meeker D, Teno JM, Lynn J, Lunney JR, Lorenz KA. Symptom trends in the last year of life from 1998 to 2010: a cohort study. Ann Intern Med. 2015 Feb 3;162(3):175-83. doi: 10.7326/M13-1609. PMID 25643305
- [Result] Bee PE, Barnes P, Luker KA. A systematic review of informal caregivers' needs in providing home-based end-of-life care to people with cancer. J Clin Nurs. 2009 May;18(10):1379-93. doi: 10.1111/j.1365-2702.2008.02405.x. Epub 2009 Apr 8. PMID 18624779
- [Result] Mayahara M, Foreman MD, Wilbur J, Paice JA, Fogg LF. Effect of hospice nonprofessional caregiver barriers to pain management on adherence to analgesic administration recommendations and patient outcomes. Pain Manag Nurs. 2015 Jun;16(3):249-56. doi: 10.1016/j.pmn.2014.07.001. Epub 2014 Nov 27. PMID 25434499
- [Result] Chi NC, Demiris G. Family Caregivers' Pain Management in End-of-Life Care: A Systematic Review. Am J Hosp Palliat Care. 2017 Jun;34(5):470-485. doi: 10.1177/1049909116637359. Epub 2016 Mar 14. PMID 26975303
- [Result] Letizia M, Creech S, Norton E, Shanahan M, Hedges L. Barriers to caregiver administration of pain medication in hospice care. J Pain Symptom Manage. 2004 Feb;27(2):114-24. doi: 10.1016/j.jpainsymman.2003.06.008. PMID 15157035
- [Result] Wilkie DJ, Kim YO, Suarez ML, Dauw CM, Stapleton SJ, Gorman G, Storfjell J, Zhao Z. Extending computer technology to hospice research: interactive pentablet measurement of symptoms by hospice cancer patients in their homes. J Palliat Med. 2009 Jul;12(7):599-602. doi: 10.1089/jpm.2009.0006. PMID 19594343
- [Result] Lind L, Karlsson D, Fridlund B. Patients' use of digital pens for pain assessment in advanced palliative home healthcare. Int J Med Inform. 2008 Feb;77(2):129-36. doi: 10.1016/j.ijmedinf.2007.01.013. Epub 2007 Mar 23. PMID 17363323
- [Result] Mayahara M, Wilbur J, O'Mahony S, Breitenstein S. E-Pain Reporter: A Digital Pain and Analgesic Diary for Home Hospice Care. J Palliat Care. 2017 Apr;32(2):77-84. doi: 10.1177/0825859717722466. Epub 2017 Sep 4. PMID 28868960
- [Result] Ward S, Donovan H, Gunnarsdottir S, Serlin RC, Shapiro GR, Hughes S. A randomized trial of a representational intervention to decrease cancer pain (RIDcancerPain). Health Psychol. 2008 Jan;27(1):59-67. doi: 10.1037/0278-6133.27.1.59. PMID 18230015
- [Result] Kutner JS, Kassner CT, Nowels DE. Symptom burden at the end of life: hospice providers' perceptions. J Pain Symptom Manage. 2001 Jun;21(6):473-80. doi: 10.1016/s0885-3924(01)00281-0. PMID 11397605
- [Result] Wilkie DJ, Ezenwa MO, Yao Y, Gill A, Hipp T, Shea R, Miller J, Carrasco J, Shuey D, Zhao Z, Angulo V, Suarez ML, McCurry T, Martin J, Molokie RE, Wang ZW. Pain Intensity and Misconceptions Among Hospice Patients With Cancer and Their Caregivers: Status After 2 Decades. Am J Hosp Palliat Care. 2017 May;34(4):318-324. doi: 10.1177/1049909116639612. Epub 2016 Mar 22. PMID 27006391
- [Result] Romem A, Tom SE, Beauchene M, Babington L, Scharf SM, Romem A. Pain management at the end of life: A comparative study of cancer, dementia, and chronic obstructive pulmonary disease patients. Palliat Med. 2015 May;29(5):464-9. doi: 10.1177/0269216315570411. Epub 2015 Feb 13. PMID 25680377
- [Result] Dawson R, Sellers DE, Spross JA, Jablonski ES, Hoyer DR, Solomon MZ. Do patients' beliefs act as barriers to effective pain management behaviors and outcomes in patients with cancer-related or noncancer-related pain? Oncol Nurs Forum. 2005 Mar 5;32(2):363-74. doi: 10.1188/05.ONF.363-374. PMID 15759073
- [Result] Zeppetella G, O'Doherty CA, Collins S. Prevalence and characteristics of breakthrough pain in patients with non-malignant terminal disease admitted to a hospice. Palliat Med. 2001 May;15(3):243-6. doi: 10.1191/026921601678576220. PMID 11407195
- [Result] Harris P, Wong E, Farrington S, Craig TR, Harrold JK, Oldanie B, Teno JM, Casarett DJ. Patterns of functional decline in hospice: what can individuals and their families expect? J Am Geriatr Soc. 2013 Mar;61(3):413-7. doi: 10.1111/jgs.12144. Epub 2013 Jan 24. PMID 23347201
- [Result] Kelley M, Demiris G, Nguyen H, Oliver DP, Wittenberg-Lyles E. Informal hospice caregiver pain management concerns: a qualitative study. Palliat Med. 2013 Jul;27(7):673-82. doi: 10.1177/0269216313483660. Epub 2013 Apr 23. PMID 23612959
- [Result] Mor V, Teno JM. Regulating and Paying for Hospice and Palliative Care: Reflections on the Medicare Hospice Benefit. J Health Polit Policy Law. 2016 Aug;41(4):697-716. doi: 10.1215/03616878-3620893. Epub 2016 Apr 28. PMID 27127256
- [Result] Koller A, Miaskowski C, De Geest S, Opitz O, Spichiger E. A systematic evaluation of content, structure, and efficacy of interventions to improve patients' self-management of cancer pain. J Pain Symptom Manage. 2012 Aug;44(2):264-84. doi: 10.1016/j.jpainsymman.2011.08.015. PMID 22871509
- [Result] Tse MM, Wong AC, Ng HN, Lee HY, Chong MH, Leung WY. The effect of a pain management program on patients with cancer pain. Cancer Nurs. 2012 Nov-Dec;35(6):438-46. doi: 10.1097/NCC.0b013e3182360730. PMID 22228392
- [Result] Nkhoma K, Seymour J, Arthur A. An Educational Intervention to Reduce Pain and Improve Pain Management for Malawian People Living With HIV/AIDS and Their Family Carers: A Randomized Controlled Trial. J Pain Symptom Manage. 2015 Jul;50(1):80-90.e4. doi: 10.1016/j.jpainsymman.2015.01.011. Epub 2015 Feb 7. PMID 25666517
- [Result] Cagle JG, Zimmerman S, Cohen LW, Porter LS, Hanson LC, Reed D. EMPOWER: an intervention to address barriers to pain management in hospice. J Pain Symptom Manage. 2015 Jan;49(1):1-12. doi: 10.1016/j.jpainsymman.2014.05.007. Epub 2014 May 28. PMID 24880000
- [Result] Capewell C, Gregory W, Closs S, Bennett M. Brief DVD-based educational intervention for patients with cancer pain: feasibility study. Palliat Med. 2010 Sep;24(6):616-22. doi: 10.1177/0269216310371704. Epub 2010 Jun 17. PMID 20558433
- [Result] Parker Oliver D, Demiris G, Washington K, Kruse RL, Petroski G. Hospice Family Caregiver Involvement in Care Plan Meetings: A Mixed-Methods Randomized Controlled Trial. Am J Hosp Palliat Care. 2017 Nov;34(9):849-859. doi: 10.1177/1049909116661816. Epub 2016 Jul 27. PMID 27465403
- [Result] Oliver DP, Wittenberg-Lyles E, Washington K, Kruse RL, Albright DL, Baldwin PK, Boxer A, Demiris G. Hospice caregivers' experiences with pain management: "I'm not a doctor, and I don't know if I helped her go faster or slower". J Pain Symptom Manage. 2013 Dec;46(6):846-58. doi: 10.1016/j.jpainsymman.2013.02.011. Epub 2013 May 31. PMID 23731855
- [Result] Besse KT, Faber-te Boveldt ND, Janssen GH, Vernooij-Dassen M, Vissers KC, Engels Y. Pain Assessment with Short Message Service and Interactive Voice Response in Outpatients with Cancer and Pain: A Feasibility Study. Pain Pract. 2016 Mar;16(3):320-6. doi: 10.1111/papr.12278. Epub 2015 Jan 12. PMID 25581306
- [Result] Wilkie DJ, Judge MK, Berry DL, Dell J, Zong S, Gilespie R. Usability of a computerized PAINReportIt in the general public with pain and people with cancer pain. J Pain Symptom Manage. 2003 Mar;25(3):213-24. doi: 10.1016/s0885-3924(02)00638-3. PMID 12614956
- [Result] Mayahara M, Wilbur J, Fogg L, Breitenstein SM, Miller AM. Feasibility of e-Pain Reporter: A Digital Pain Management Tool for Informal Caregivers in Home Hospice. J Hosp Palliat Nurs. 2019 Jun;21(3):193-199. doi: 10.1097/NJH.0000000000000548. PMID 31045994
- [Result] Gunnarsdottir S, Serlin RC, Ward S. Patient-related barriers to pain management: the Icelandic Barriers Questionnaire II. J Pain Symptom Manage. 2005 Mar;29(3):273-85. doi: 10.1016/j.jpainsymman.2004.06.015. PMID 15781178
- [Result] Lind L, Karlsson D. A system for symptom assessment in advanced palliative home healthcare using digital pens. Med Inform Internet Med. 2004 Sep-Dec;29(3-4):199-210. doi: 10.1080/14639230400005966. PMID 15742987
- [Result] Ugalde A, Krishnasamy M, Schofield P. Development of an instrument to measure self-efficacy in caregivers of people with advanced cancer. Psychooncology. 2013 Jun;22(6):1428-34. doi: 10.1002/pon.3160. Epub 2012 Sep 3. PMID 22941754
- [Result] Mayahara M, Fogg L. Examination and Analysis of After-Hours Calls in Hospice. Am J Hosp Palliat Care. 2020 May;37(5):324-328. doi: 10.1177/1049909119900377. Epub 2020 Jan 30. PMID 31996017
- [Result] Baik D, Russell D, Jordan L, Dooley F, Bowles KH, Masterson Creber RM. Using the Palliative Performance Scale to Estimate Survival for Patients at the End of Life: A Systematic Review of the Literature. J Palliat Med. 2018 Nov;21(11):1651-1661. doi: 10.1089/jpm.2018.0141. Epub 2018 Aug 21. PMID 30129809
- [Result] Lau F, Maida V, Downing M, Lesperance M, Karlson N, Kuziemsky C. Use of the Palliative Performance Scale (PPS) for end-of-life prognostication in a palliative medicine consultation service. J Pain Symptom Manage. 2009 Jun;37(6):965-72. doi: 10.1016/j.jpainsymman.2008.08.003. Epub 2009 Feb 20. PMID 19232892
- [Result] Ward SE, Serlin RC, Donovan HS, Ameringer SW, Hughes S, Pe-Romashko K, Wang KK. A randomized trial of a representational intervention for cancer pain: does targeting the dyad make a difference? Health Psychol. 2009 Sep;28(5):588-597. doi: 10.1037/a0015216. PMID 19751085
- [Result] Bonsignore L, Bloom N, Steinhauser K, Nichols R, Allen T, Twaddle M, Bull J. Evaluating the Feasibility and Acceptability of a Telehealth Program in a Rural Palliative Care Population: TapCloud for Palliative Care. J Pain Symptom Manage. 2018 Jul;56(1):7-14. doi: 10.1016/j.jpainsymman.2018.03.013. Epub 2018 Mar 16. PMID 29551433
- [Result] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Result] Chou R, Gordon DB, de Leon-Casasola OA, Rosenberg JM, Bickler S, Brennan T, Carter T, Cassidy CL, Chittenden EH, Degenhardt E, Griffith S, Manworren R, McCarberg B, Montgomery R, Murphy J, Perkal MF, Suresh S, Sluka K, Strassels S, Thirlby R, Viscusi E, Walco GA, Warner L, Weisman SJ, Wu CL. Management of Postoperative Pain: A Clinical Practice Guideline From the American Pain Society, the American Society of Regional Anesthesia and Pain Medicine, and the American Society of Anesthesiologists' Committee on Regional Anesthesia, Executive Committee, and Administrative Council. J Pain. 2016 Feb;17(2):131-57. doi: 10.1016/j.jpain.2015.12.008. PMID 26827847
- [Result] Bellg AJ, Borrelli B, Resnick B, Hecht J, Minicucci DS, Ory M, Ogedegbe G, Orwig D, Ernst D, Czajkowski S; Treatment Fidelity Workgroup of the NIH Behavior Change Consortium. Enhancing treatment fidelity in health behavior change studies: best practices and recommendations from the NIH Behavior Change Consortium. Health Psychol. 2004 Sep;23(5):443-51. doi: 10.1037/0278-6133.23.5.443. PMID 15367063
- [Result] Polit DF, Beck CT. The content validity index: are you sure you know what's being reported? Critique and recommendations. Res Nurs Health. 2006 Oct;29(5):489-97. doi: 10.1002/nur.20147. PMID 16977646
- [Result] McMillan SC, Moody LE. Hospice patient and caregiver congruence in reporting patients' symptom intensity. Cancer Nurs. 2003 Apr;26(2):113-8. doi: 10.1097/00002820-200304000-00004. PMID 12660560
- [Result] Morisky DE, Green LW, Levine DM. Concurrent and predictive validity of a self-reported measure of medication adherence. Med Care. 1986 Jan;24(1):67-74. doi: 10.1097/00005650-198601000-00007. PMID 3945130
- [Result] Hsieh HF, Shannon SE. Three approaches to qualitative content analysis. Qual Health Res. 2005 Nov;15(9):1277-88. doi: 10.1177/1049732305276687. PMID 16204405
- [Result] Mayahara M, Miller AM, O'Mahony S. Components of the Advance Care Planning Process in the Nursing Home Setting. J Hosp Palliat Nurs. 2018 Feb;20(1):95-102. doi: 10.1097/NJH.0000000000000414. PMID 30063620
- [Result] Graneheim UH, Lundman B. Qualitative content analysis in nursing research: concepts, procedures and measures to achieve trustworthiness. Nurse Educ Today. 2004 Feb;24(2):105-12. doi: 10.1016/j.nedt.2003.10.001. PMID 14769454
- [Derived] Mayahara M, Wilbur J, Fogg L, Houlihan MC, Oliver DP, Benson JJ, Miller AM. The e-PainSupport Digital Application for Assessing Pain and Pain Management in Home Hospice: A Randomized Controlled Trial. West J Nurs Res. 2025 Aug;47(8):708-719. doi: 10.1177/01939459251338392. Epub 2025 Jun 10. PMID 40495339